CLINICAL TRIAL: NCT04951232
Title: Cinepazide Maleate Injection in the Treatment of Acute Ischemic Stroke A Blind, Multicenter, Placebo-controlled Clinical Confirmatory Study.
Brief Title: Clinical Study of Cinepazide Maleate Injection in the Treatment of Acute Ischemic Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Collaborators: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D2016058
Record Dates: First submitted 2021-06-27; First posted 2021-07-06 (Actual); Last update posted 2021-07-06 (Actual); Status verified 2021-06

CONDITIONS: Stroke, Ischemic
MeSH Terms: conditions — Ischemic Stroke | interventions — cinepazide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (cinnarizide maleate injection group) (Experimental)
  Interventions: Drug: Cinepazide Maleate
- control group (placebo group) (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Cinepazide Maleate — The experimental group: guipiprazitel maleate injection (klingo): 320mg (4), dissolved in 500ml of normal saline, and injected in a medium vein at a rate of 100ml/h, once a day, and administered for 14 days.
  Arms: Test group (cinnarizide maleate injection group)
Other: Placebo — Placebo: 4 pieces, dissolved in normal saline 500ml, intravenous drip, the speed is 100ml / h, once a day, continuous administration for 14 days
  Arms: control group (placebo group)

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled, parallel controlled, post marketing confirmatory clinical trial in Chinese patients with acute ischemic stroke. Objective to evaluate the efficacy and safety of cinepazide maleate injection compared with placebo in the treatment of patients with acute ischemic stroke.

DETAILED DESCRIPTION:
The target population of this study is patients with acute ischemic stroke within 48 hours. All potential participants must provide informed consent, and those who provide informed consent will enter the screening (- 48 ~ 0h), and the screening qualification will be evaluated according to the inclusion criteria. The eligible subjects will enter the treatment period (day 1-14) and will be randomly assigned to the experimental group (cinepazide maleate injection group) or the control group (placebo group).

During the treatment period, all subjects will receive cinepazide maleate injection or placebo by intravenous drip at the rate of 100ml / h, once a day for 14 consecutive days. During the treatment, all subjects need to receive basic treatment: citicoline sodium injection 0.5g, dissolved in 5% glucose injection or normal saline 250ml, intravenous drip slowly, once a day, continuous administration for 10 days. According to the Chinese guidelines for the diagnosis and treatment of acute ischemic stroke (2014), the patients were given antihypertensive, hypoglycemic, lipid-lowering, anticoagulant or mannitol. All subjects were not allowed to receive interventional therapy, thrombolysis (such as rtPA and urokinase), defibrillator, any platelet inhibitor except aspirin and clopidogrel, other cerebrovascular dilators (such as cinnarizine, flunarizine, nicardipine and nimodipine), other neuroprotective agents (except citicoline) during the whole trial period After the end of the treatment period (the 14th day), the subjects will enter the follow-up period (the 15th-90th day).

During the follow-up period, subjects need to be followed up twice (30th day) ± 2 days, 90th day ± 3 days).

ELIGIBILITY:
Inclusion Criteria:

* 1. 18-80 years old (contains 18 and 80 years), with no limit for both sexes; 2. Acute internal carotid artery was diagnosed according to the Chinese guidelines for the diagnosis and treatment of acute ischemic stroke (2014) Cerebral infarction of the arterial system (anterior circulation), well after first onset or last onset (MRS score 0-1) patients; 3. Onset ≤ 48 hours (onset to randomization within 48 hours); 4. 5 points ≤ NIHSS ≤ 25 at presentation; 5. Informed consent was signed by the patients or their legal surrogates.

Exclusion Criteria:

* 1. Patients with recurrent cerebral infarction with pre Mrs score ≥ 2 at this time; 2. Cranial CT suggestive of intracranial haemorrhagic disease (e.g Intracranial hematoma, intraventricular hemorrhage, subarachnoid hemorrhage, etc.); 3. Cerebral infarction with impaired consciousness (NIHSS score of 1A items ≥ 1), transient ischemic attack Zuo, cerebral arteritis, brain tumor, brain trauma, intracranial infection, cerebral parasite disease patients; 4. Patients who have undergone or require interventional, thrombolytic, and defibrillation therapy after this episode; 5. History or evidence of any one of the following diseases during the screening period:

  * poorly controlled hypertension with systolic blood pressure ≥ 200mmhg or diastolic blood pressure ≥ 110mmhg during screening period;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2016-07-04 (Actual); Primary Completion 2017-01-06 (Actual); Study Completion 2017-01-06 (Actual)

PRIMARY OUTCOMES:
score of modified Rankin Scale(MRS) | at day 90
  proportion of subjects with a modified Rankin Scale (MRS) ≤ 2

SECONDARY OUTCOMES:
ability of daily life | at day 90
  the score of Barth index(BI)

CONTACTS AND LOCATIONS:
Overall Officials: Dongsheng Fan, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No